CLINICAL TRIAL: NCT00089986
Title: A Prospective, Randomized, Double-blind, Placebo Controlled, Dose Ranging, Multi-Center Study of the Safety and Efficacy of Three Days Continuous Intravenous Infusion of GR270773 in the Treatment of Suspected or Confirmed Gram-negative Severe Sepsis in Adults
Brief Title: GR270773 In The Treatment Of Suspected Or Confirmed Gram-Negative Severe Sepsis In Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: EMD20001
Record Dates: First submitted 2004-08-18; First posted 2004-08-23 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Sepsis
Keywords: severe sepsis; septic shock; Gram-negative infection; phospholipid emulsion
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intravenous GR270773- Phospholipid Emulsion
Other: Placebo
  Other Names: Matched placebo infusion

SUMMARY:
The primary objective is to estimate the size of the GR270773 treatment effect on 28-day all-cause mortality for two doses of GR270773 versus placebo in adult subjects with suspected or confirmed Gram-negative severe sepsis. GR270773 will be administered as a three-day continuous intravenous infusion.

ELIGIBILITY:
Inclusion criteria:

* Receiving parenteral antibiotic therapy for a suspected or confirmed Gram-negative infection.
* Have at least one new hypoperfusion abnormality or at least one new onset organ failure resulting from the current septic episode.
* Must be available and able to receive the first dose of study medication no more than 12 hours after the confirmation of a new hypoperfusion abnormality or new onset organ failure and within 36 hours after the initiation of new parenteral antibacterial therapy for the suspected or confirmed Gram-negative infection believed to be responsible for this episode of sepsis.

Exclusion criteria:

* Subject is unlikely to remain in hospital for a minimum of three days (72 hours) following enrollment.
* Subject has neutropenia (e.g., subject recently receiving cytotoxic chemotherapy with absolute neutrophil count <500/mcL or expected to decline to <500/mcL in the next 3 days).
* Subject has known active hemolytic disease, immune hemolytic anemias, hemoglobinopathies (sickle cell anemia and thalassemia major).
* Subject has a known bone marrow disorder of inadequate red cell production (eg, aplastic anemia, myelodysplasia).
* Subject is at increased risk of complications from GR270773-related hemolysis due to the inability to increase cardiac function sufficiently to meet the demands for oxygen delivery.
* Subject has a baseline hemoglobin (measured after adequate volume resuscitation) <9.0 g/dL (5.59 mmol/L).
* Subject is currently being treated with XIGRIS (Drotrecogin alfa (activated)) or its use is considered imminent (ie., a decision to treat with XIGRIS has been made).
* Subject has a history of allergic reaction to eggs (or egg products), soybeans, INTRALIPID, or any component of GR270773.
* Subject has been designated as 'not full support do not resuscitate' (DNR), or other equivalent status which prohibits the use of life supporting interventions (e.g., mechanical ventilation, dialysis/hemofiltration, or others) thereby limiting the treatment options available.

Note: Subjects with advanced directives prohibiting only chest compression (CPR) are eligible for the study.

* Subject has preexisting severe liver disease such as cirrhosis, primary biliary cirrhosis or known preexisting Child-Pugh class B or C liver dysfunction.
* Subject is moribund (a state in which death is perceived to be imminent) or has a life expectancy of less than 3 months due to an underlying disease.
* Subject is currently receiving one of the following prohibited concomitant medications; parenteral nutrition supplements containing lipid emulsions (e.g., INTRALIPID), amphotericin, liposomal amphotericin, or amphotericin B lipid complex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1415 (Actual)
Dates: Start 2004-09-01; Primary Completion 2007-04-01 (Actual); Study Completion 2007-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (305):
- United States (113):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bentonville, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Atlantis, Florida
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Rome, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Naperville, Illinois
  - GSK Investigational Site, North Chicago, Illinois
  - GSK Investigational Site, Oak Park, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, East Lansing, Michigan
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Piscataway, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Monroeville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Pawtucket, Rhode Island
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lackland Air Force Base, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Burlington, Vermont
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, Marshfield, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (5):
  - GSK Investigational Site, Villa Sarmiento-Haedo, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires
  - GSK Investigational Site, Moron-Provincia de Buenos Aires
- Australia (5):
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Footscray, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Nedlands, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- Austria (2):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- Belgium (7):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Ottignies
  - GSK Investigational Site, Yvoir
- Brazil (3):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Ribeirão Preto, São Paulo
  - GSK Investigational Site, São Paulo
- Canada (16):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (9):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Joensuu
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lappeenranta
  - GSK Investigational Site, Mikkeli
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
- France (15):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Argenteuil
  - GSK Investigational Site, Bourg-en-Bresse
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Le Chesnay
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montauban
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Michel
- Germany (34):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Greifswald, Mecklenburg-Vorpommern
  - GSK Investigational Site, Neubrandenburg, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Wismar, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Bad Berka, Thuringia
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bremen
  - GSK Investigational Site, Hamburg
- Greece (5):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari
  - GSK Investigational Site, Kifissia
  - GSK Investigational Site, Rio, Patras
  - GSK Investigational Site, Thessaloniki
- Hong Kong (4):
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
  - GSK Investigational Site, Tuen Mun, New Territories
- GSK Investigational Site, Budapest, Hungary
- India (5):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Mangalore
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Pune
- Israel (5):
  - GSK Investigational Site, Afula
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Zrifin
- GSK Investigational Site, Riga, Latvia
- Malaysia (2):
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kubang Kerian
- Netherlands (7):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Apeldoorn
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- New Zealand (3):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Tauranga
- Portugal (3):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Lisbon
- GSK Investigational Site, San Juan, Puerto Rico
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
- Russia (8):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburgh
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yekaterinburg
- Slovenia (6):
  - GSK Investigational Site, Celje
  - GSK Investigational Site, Ljubljana
  - GSK Investigational Site, Maribor
  - GSK Investigational Site, Novo Mesto
  - GSK Investigational Site, Slovenj Gradec
  - GSK Investigational Site, Šempeter Pri Novi Gorici
- South Africa (6):
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Auckland Park, Johannesburg
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, George
  - GSK Investigational Site, PO Medunsa
- GSK Investigational Site, Seoul, South Korea
- Spain (10):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Tarrasa
  - GSK Investigational Site, Terrassa
  - GSK Investigational Site, Valencia
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
- Taiwan (4):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan County
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- United Kingdom (10):
  - GSK Investigational Site, Aberdeen, Aberdeenshire
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Wigan, Lancashire
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Oxford, Oxfordshire
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Livingston, West Lothian
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 1845 participants, hospitalized with suspected or confirmed gram-negative severe sepsis, male or female >=18 years of age at 235 centers across 31 countries from 02 September 2004 to 25 June 2007.
Pre-assignment Details: A total of 1415 participant numbers were assigned during randomization process, five were duplicate randomization numbers and for other two, the participants did not provide informed consent, precluding them from enrollment. Out of 1408 participants, 29 did not receive study medication, remaining 1379 included in Intent-to-Treat (ITT) Population.
Groups:
- Placebo: Eligible participants were administered matching placebo to low-dose GR270773 or high-dose GR270773, intravenously (IV) as a loading dose infused over 2 hours (h) followed by a maintenance dose administered as a continuous infusion for 70 h, for a total treatment period of 72 h. The low placebo rate consisted of a loading dose of 0.75 milliliters per kilogram per hour (mL/kg/h) for 2 h and a maintenance dose of 0.1 mL/kg/h for 70 h. The high placebo rate consisted of a loading dose of 1.5 mL/kg/h for 2 h and a maintenance dose of 0.15 mL/kg/h for 70 h.
- Low GR270773: Eligible participants were administered low-dose GR270773 IV as a loading dose infused over 2 h followed by a maintenance dose administered as a continuous infusion for 70 h, for a total treatment period of 72 h. The study medication was administered as a sterile 100 milligrams per milliliter (mg/mL) lipid emulsion for IV administration. The low dose emulsion consisted of a loading dose of 75 milligram (mg)/kg/h which was equivalent to 0.75 mL/kg/h for 2 h and a maintenance dose of 10 mg/kg/h which was equivalent to 0.1 mL/kg/h for 70 h. The total dose was 850 mg/kg.
- High GR270773: Eligible participants were administered high-dose GR270773 IV as a loading dose infused over 2 h followed by a maintenance dose administered as a continuous infusion for 70 h, for a total treatment period of 72 h. The study medication was administered as a sterile 100 mg/mL lipid emulsion for IV administration. The high dose emulsion consisted of a loading dose of 15 mg/kg/h which was equivalent to 1.5 mL/kg/h for 2 h and a maintenance dose of 15 mg/kg/h which was equivalent to 0.15 mL/kg/h for 70 h. The total dose was 1350 mg/kg.
Period: Overall Study
Arm/Group | Placebo | Low GR270773 | High GR270773
Started | 599 | 598 | 182
Completed | 584 | 574 | 172
Not Completed | 15 | 24 | 10
Not completed — Adverse Event | 6 | 9 | 6
Not completed — Lost to Follow-up | 3 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Patient transferred to another hospital | 2 | 1 | 0
Not completed — Subject withdrew but agreed follow up | 1 | 2 | 0
Not completed — Hemohlobin stopping rule | 0 | 1 | 0
Not completed — Investigator decision to withdrew | 0 | 1 | 0
Not completed — Enrollment in another study | 0 | 1 | 0
Not completed — Family decision | 0 | 1 | 0
Not completed — Do not resuscitate (DNR) | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants were administered matching placebo to low-dose GR270773 or high-dose GR270773, IV as a loading dose infused over 2 h followed by a maintenance dose administered as a continuous infusion for 70 h, for a total treatment period of 72 h. The low placebo rate consisted of a loading dose of 0.75 mL/kg/h for 2 h and a maintenance dose of 0.1 mL/kg/h for 70 h. The high placebo rate consisted of a loading dose of 1.5 mL/kg/h for 2 h and a maintenance dose of 0.15 mL/kg/h for 70 h.
- Low GR270773: Eligible participants were administered low-dose GR270773 IV as a loading dose infused over 2 h followed by a maintenance dose administered as a continuous infusion for 70 h, for a total treatment period of 72 h. The study medication was administered as a sterile 100 mg/mL lipid emulsion for IV administration. The low dose emulsion consisted of a loading dose of 75 mg/kg/h which was equivalent to 0.75 mL/kg/h for 2 h and a maintenance dose of 10 mg/kg/h which was equivalent to 0.1 mL/kg/h for 70 h. The total dose was 850 mg/kg.
- Total: Total of all reporting groups
Arm/Group | Placebo | Low GR270773 | High GR270773 | Total
Number analyzed (Participants) | 599 | 598 | 182 | 1379
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (16.41) | 62.8 (16.27) | 64.8 (15.47) | 63.2 (16.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 239 | 80 | 573
  Male | 345 | 359 | 102 | 806
Race/Ethnicity, Customized [Number; unit: Participants]
  Arabic/North African | 7 | 6 | 1 | 14
  Black | 16 | 14 | 2 | 32
  East & South East Asian | 51 | 44 | 14 | 109
  Japanese | 3 | 3 | 0 | 6
  South Asian | 29 | 32 | 2 | 63
  White/Caucasian | 484 | 494 | 161 | 1139
  Pacific Islander | 1 | 0 | 0 | 1
  American Indian | 4 | 2 | 0 | 6
  Native Hawaiian | 2 | 0 | 0 | 2
  Missing | 2 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 28-Day All Cause Mortality
Description: Mortality was assessed by the number of participants who died between days 1 and 28. A summary of death details was given which included whether the participant died between days 1 and 28, whether the death was related sepsis, cause of death, the source of the information, and whether the cause of death was verified by a death record. Participants who had withdrawn from study and all study assessments and for whom survival at day 28 could not be confirmed was treated as deaths for the primary endpoint. The difference in all-cause 28-day mortality rates for each treatment group versus the placebo group in the ITT Population was calculated as placebo - treatment.
Time Frame: Day 1 (post-infusion) up to Day 28 Follow-up
Population: ITT Population was defined as all randomized participants from all three stages who receive any study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Low GR270773 | High GR270773
Number analyzed (Participants) | 599 | 598 | 182
Percentage of participants | 26.9 | 25.8 | 31.3
Statistical Analysis 1: Comparison: Placebo vs Low GR270773; Test type: Superiority or Other; p = 0.329, Chi-squared; Rate difference = 1.1, 90% CI 1-sided [lower limit -2.1]
Statistical Analysis 2: Comparison: Placebo vs High GR270773; Test type: Superiority or Other; p = 0.879, Chi-squared; Rate Difference = -4.4, 90% CI 1-sided [lower limit -9.4]

2. Secondary Outcome: Number of Participants With New Onset Organ Failure, Regardless of Cause, Occurring During the 28 Days Post Enrollment in an Organ Not in Failure at Enrolment
Description: The new onset organ failure was defined as first time each of the following criteria were met after start of study medication up to Day 28. Respiratory failure: defined by requiring mechanical ventilation not less than 24 hours due to surgery. Renal failure: defined by requiring the initiation of hemodialysis or hemofiltration. Coagulopathy: defined by disseminated intravascular coagulation (DIC) requiring transfusion with platelets or fresh frozen plasma or anticoagulant therapy. Cardiovascular failure: defined by sustained hypotension requiring vasopressor support of dopamine >5 microgram per kilogram per minute (µg/kg/min), epinephrine, norepinephrine, phenylephrine or vasopressin at any dose if used to increase blood pressure for >=6 continuous h. Analysis was done treating the death as a new onset organ failure (counted in both the numerator and denominator).
Time Frame: Baseline (Day 1, pre-infusion) up to Day 28 Follow-up
Population: ITT Population. Organ failure occurring during the 28 days post-enrollment that was not in failure at enrollment. Subjects who die prior to observing a new organ failure are counted as a failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low GR270773 | High GR270773
Number analyzed (Participants) | 599 | 598 | 182
Participants | 122 | 157 | 57

3. Secondary Outcome: Number of Participants With New Onset Organ Failure of Respiratory Failure, Cardiovascular Failure, Renal Failure and Coagulopathy, Regardless of Cause, Occurring During the 28 Days Post Enrollment in an Organ Not in Failure at Enrollment
Description: Respiratory failure: defined by requiring mechanical ventilation not less than 24 hours due to surgery. Renal failure: defined by requiring the initiation of hemodialysis or hemofiltration. Coagulopathy: defined by disseminated intravascular coagulation (DIC) requiring transfusion with platelets or fresh frozen plasma or anticoagulant therapy. Cardiovascular failure: defined by sustained hypotension requiring vasopressor support of dopamine >5 microgram per kilogram per minute (µg/kg/min), epinephrine, norepinephrine, phenylephrine or vasopressin at any dose if used to increase blood pressure for >=6 continuous h. For each organ failure type and the number of new onset organ failures per participants for each organ failure type, the denominator only included participants who did not have that type of organ failure at Baseline. At Baseline a participant could enter the study with a type of organ failure, that type of failure was not reported as a new onset organ failure.
Time Frame: Baseline (Day 1, pre-infusion) up to Day 28 Follow up
Population: ITT Population. Organ failure occurring during the 28 days post-enrollment that was not in failure at enrollment. Participants who died prior to observing a new failure are excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low GR270773 | High GR270773
Number analyzed (Participants) | 599 | 598 | 182
Participants
  Respiratory failure, n= 297, 333, 99 | 50 | 61 | 23
  Cardiovascular failure, n= 150, 161, 43 | 33 | 48 | 15
  Renal failure, n= 460, 474, 138 | 40 | 47 | 22
  Coagulopathy, n= 344, 355, 107 | 36 | 41 | 16

4. Secondary Outcome: Assessment of Safety/Tolerability by Determining the Number of Participants With Any Adverse Events (AE), Serious Adverse Events (SAE) and Fatal SAE
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition or common toxicity criteria (CTC) grade 4 laboratory abnormalities of national cancer institute not associated with the underlying sepsis unless more severe than expected for the participants condition.
Time Frame: Day 1 (pre-infusion) up to Day 28 Follow-up
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low GR270773 | High GR270773
Number analyzed (Participants) | 599 | 598 | 182
Participants
  Any AE | 423 | 442 | 144
  Any SAE | 213 | 235 | 77
  Any fatal SAE | 85 | 70 | 33

ADVERSE EVENTS:
Time Frame: AE and SAE were collected from Baseline (Day 1, pre-infusion) to Day 28 Follow-up
Description: ITT Population was used which was defined as all randomized participants from all three stages who receive any study drug.
Arm/Group | Placebo | Low GR270773 | High GR270773
All-Cause Mortality (participants affected / at risk) | 85/599 | 70/598 | 33/182
Serious Adverse Events (participants affected / at risk) | 213/599 | 235/598 | 77/182
Other Adverse Events (participants affected / at risk) | 160/599 | 183/598 | 60/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=599) | Low GR270773 (N=598) | High GR270773 (N=182)
Metabolic acidosis (Metabolism and nutrition disorders) | 49 | 61 | 23
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 10 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 46 | 42 | 17
Atrial fibrillation (Cardiac disorders) | 3 | 6 | 1
Myocardial infarction (Cardiac disorders) | 4 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 3 | 3
Ventricular tachycardia (Cardiac disorders) | 4 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 3 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 2 | 0
Torsade de pointes (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Mental impairment (Nervous system disorders) | 38 | 38 | 12
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 1
Brain oedema (Nervous system disorders) | 1 | 2 | 1
Anoxic encephalopathy (Nervous system disorders) | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Encephalitis (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hypoxic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 20 | 25 | 15
Cholangitis (Hepatobiliary disorders) | 1 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 2 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 4 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 3 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic duct obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Lipase increased (Investigations) | 7 | 10 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 3 | 0
Haemoglobin decreased (Investigations) | 2 | 2 | 0
Hepatic enzyme increased (Investigations) | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0
Blood amylase increased (Investigations) | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Carbon dioxide decreased (Investigations) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Cardiac output decreased (Investigations) | 1 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0
Myelocyte present (Investigations) | 0 | 1 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 2
Septic shock (Infections and infestations) | 6 | 2 | 0
Sepsis (Infections and infestations) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Wound infection (Infections and infestations) | 1 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Citrobacter sepsis (Infections and infestations) | 0 | 0 | 1
Colitis pseudomembranous (Infections and infestations) | 0 | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0
Extradural abscess (Infections and infestations) | 1 | 0 | 0
Fungaemia (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0
Perinephric abscess (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemopneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 8 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2 | 0
Coombs negative haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Red blood cell abnormality (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 2 | 3
Deep vein thrombosis (Vascular disorders) | 2 | 2 | 0
Shock haemorrhagic (Vascular disorders) | 3 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0
Heart injury (Injury, poisoning and procedural complications) | 3 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 2 | 0
Graft complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 2 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0
Failure to anastomose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Bladder distension (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 1
Multi-organ failure (General disorders) | 3 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 1
Cardiac death (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Hyperpyrexia (General disorders) | 0 | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=599) | Low GR270773 (N=598) | High GR270773 (N=182)
Anaemia (Blood and lymphatic system disorders) | 76 | 87 | 28
Diarrhoea (Gastrointestinal disorders) | 33 | 50 | 28
Nausea (Gastrointestinal disorders) | 25 | 31 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 51 | 53 | 16
Atrial fibrillation (Cardiac disorders) | 44 | 41 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.